CLINICAL TRIAL: NCT00316862
Title: A Phase II Trial of Preoperative Irinotecan, Cisplatin and Radiation in Esophageal Cancer
Brief Title: Cisplatin, Irinotecan, and Radiation Therapy in Treating Patients With Esophageal Cancer or Gastroesophageal Junction Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-80302; CDR0000468495 (Registry Identifier: NCI Physician Data Query); NCI-2009-00491 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; stage II esophageal cancer; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Irinotecan; Radiotherapy; Radiation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy, chemoradiotherapy, surgery) (Experimental): INDUCTION CHEMOTHERAPY (COURSES 1-2): Patients receive cisplatin intravenously (IV) over 30 minutes and irinotecan hydrochloride IV over 30-90 minutes on days 1 and 8 of courses 1 and 2. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  CHEMORADIOTHERAPY (COURSES 3-4): Beginning 2 weeks after completion of induction chemotherapy, patients receive cisplatin and irinotecan hydrochloride as in induction chemotherapy on days 1 and 8 of courses 3 and 4 and undergo radiotherapy daily 5 days a week in course 3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  SURGERY: Approximately 4-8 weeks after completion of chemoradiotherapy, patients undergo surgery to remove the tumor.
  Interventions: Drug: cisplatin; Drug: irinotecan hydrochloride; Procedure: therapeutic conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — Given IV
Drug: irinotecan hydrochloride — Given IV
Procedure: therapeutic conventional surgery — Undergo Surgery
Radiation: radiation therapy — Undergo radiation
  Other Names: irradiation, radiotherapy, therapy, radiation

SUMMARY:
This phase II trial studies how well giving cisplatin and irinotecan hydrochloride together with radiation therapy works in treating patients with esophageal cancer or gastroesophageal junction cancer that can be removed by surgery. Drugs used in chemotherapy, such as cisplatin and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the pathologic complete response rate in patients with surgically resectable esophageal cancer treated pre-operatively with induction chemotherapy with weekly cisplatin and irinotecan (irinotecan hydrochloride) followed by concurrent cisplatin/irinotecan and radiation therapy.

SECONDARY OBJECTIVES:

I. To evaluate potential response or progression of disease during induction chemotherapy with positron emission tomography (PET) scan.

II. To evaluate the toxicity and tolerability of therapy, including surgical morbidity and mortality.

III. To determine the overall survival, disease free survival, and pattern of failure.

OUTLINE:

INDUCTION CHEMOTHERAPY (COURSES 1-2): Patients receive cisplatin intravenously (IV) over 30 minutes and irinotecan hydrochloride IV over 30-90 minutes on days 1 and 8 of courses 1 and 2. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

CHEMORADIOTHERAPY (COURSES 3-4): Beginning 2 weeks after completion of induction chemotherapy, patients receive cisplatin and irinotecan hydrochloride as in induction chemotherapy on days 1 and 8 of courses 3 and 4 and undergo radiotherapy daily 5 days a week in course 3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

SURGERY: Approximately 4-8 weeks after completion of chemoradiotherapy, patients undergo surgery to remove the tumor.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
* Histologically or cytologically confirmed adenocarcinoma, poorly differentiated carcinoma, or carcinoma not otherwise specified, of the esophagus or gastroesophageal junction; biopsy or cytology of the primary tumor, or of involved regional lymph nodes, is acceptable
* Tumors must be TNM stage T2-4, N0-1, M0 as determined by pretreatment endoscopic ultrasound; T1 tumors are eligible if they are T1, N1, M0; regional thoracic lymph node involvement (N1) is permitted
* Disease must be clinically limited to the esophagus or gastroesophageal junction; if the tumor extends below the gastroesophageal junction into the proximal stomach, 50% of the tumor must involve the distal esophagus or gastroesophageal junction; adenocarcinomas of the distal esophagus would therefore include tumors of the distal esophagus, or Siewert type I according to the Siewert classification, and tumors of the gastroesophageal junction which involve equally both the distal esophagus and proximal stomach, or Siewert type II; tumor must be surgically resectable

  * No TIS (in-situ carcinoma) and tumors determined to be T1N0 following endoscopic ultrasound
  * No clinical involvement on endoscopic ultrasound (EUS), computed tomography (CT) scan, or PET scan of supraclavicular or celiac lymph node involvement (stage IVa, T any N any M1a) unless this is proven to be a false positive by an appropriate biopsy
  * No patients with cervical esophageal tumors, or gastric cancers with minor involvement of the gastroesophageal junction or distal esophagus
  * No patients with tracheoesophageal fistulas
* Patients with evidence of metastatic disease are not eligible; this includes:

  * Positive malignant cytology of the pleura, pericardium or peritoneum
  * Radiographic evidence of distance organ involvement including lung, liver, bone, or brain
* No prior chemotherapy or radiotherapy is permitted; patients must be at least 4 weeks since major surgery, or must have recovered from the effects of minor surgery (laparoscopy, thoracoscopy)
* No prior malignancies (other than basal cell/squamous carcinoma of the skin, in-situ cervical carcinoma, or superficial transitional cell bladder carcinoma) are permitted unless diagnosed and/or treated >= 3 years before registration and without evidence of recurrence
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* No evidence of recurrent laryngeal nerve or phrenic nerve paralysis
* No known Gilbert's disease
* No clinically significant hearing loss; audiograms should be done in patients in which they are clinically indicated
* No history of active seizure disorder; no ongoing treatment with phenytoin, phenobarbital, or other antiepileptic medication; patients who are receiving valproic acid are eligible
* No New York Heart Association class III or IV heart disease; no angina or myocardial infarction within the last 6 months

Inclusion Criteria:

* No history of clinically significant ventricular arrhythmia requiring ongoing medication with antiarrhythmics
* Absolute neutrophil count (ANC) >= 1,500/ul
* Platelet count >= 100,000/ul
* Hemoglobin >= 9 gm/dl
* Serum creatinine =< upper limit of normal (ULN)
* Total serum bilirubin =< 1.5 mg/dl
* Forced expiratory volume in 1 second (FEV-1) >= 1.2 liters OR >= 35% of normal as a value that is indexed to body size
* Pulmonary function tests (PFT) >= 1.2 liters OR >= 35% of normal as a value that is indexed to body size

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (24):
- United States (24):
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2006 and August 2011, 82 participants were recruited to this study.
Groups:
- Treatment (Chemotherapy, Chemoradiotherapy, Surgery): INDUCTION CHEMOTHERAPY (COURSES 1-2): Patients receive cisplatin 30 mg/m^2 intravenously (IV) over 30 minutes and irinotecan hydrochloride 65 mg/m^2 IV over 30-90 minutes on days 1 and 8 of courses 1 and 2. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  CHEMORADIOTHERAPY (COURSES 3-4): Beginning 2 weeks after completion of induction chemotherapy, patients receive cisplatin and irinotecan hydrochloride as in induction chemotherapy on days 1 and 8 of courses 3 and 4 and undergo radiotherapy daily 5 days a week in course 3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  SURGERY: Approximately 4-8 weeks after completion of chemoradiotherapy, patients undergo surgery to remove the tumor.
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Chemoradiotherapy, Surgery)
Started | 82
Completed | 82
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Chemoradiotherapy, Surgery)
Number analyzed (Participants) | 82
Age, Continuous [Median (Full Range); unit: years] | 62.2 [37.3 to 85.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 77
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 77
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 82

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Adenocarcinoma Achieving a Pathologic Complete Response (CR) After Surgery
Description: A pathological complete response is defined as no tumor found on pathology review at surgery in all resected lymph nodes and tissue. All tissues sampled must have NO viable tumor
Time Frame: Up to 5 years
Population: 27 participants with adenocarcinoma were recruited and evaluated for the primary outcome per protocol design.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Chemotherapy, Chemoradiotherapy, Surgery)
Number analyzed (Participants) | 27
percentage of participants | 19 [6 to 38]

2. Secondary Outcome: Utility of Early PET Imaging in Predicting Response to Treatment
Time Frame: Up to 55 days
Reporting Status: Not Posted

3. Secondary Outcome: Disease-free Survival
Time Frame: Up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Patterns of Failure
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Proportion of Patients Experiencing Grade 3 or Greater Pneumonitis or Esophagitis
Description: Proportion of patients experiencing grade 3 or greater pneumonitis or esophagitis, deemed at least possibly related to treatment graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Time Frame: Up to 5 years
Population: 1 participant was not evaluated for adverse events.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Chemotherapy, Chemoradiotherapy, Surgery)
Number analyzed (Participants) | 81
percentage of participants
  Pneumonitis | 0
  Esophagitis | 5

7. Secondary Outcome: Proportion of Patients Experiencing Grade 3 or Greater Hematologic and Non-hematologic Toxicity
Description: Proportion of patients experiencing grade 3 or greater hematologic and non-hematologic toxicity, deemed as at least possibly related to treatment, graded using the NCI CTCAE version 3.0
Time Frame: Up to 5 years
Population: 1 participant was not evaluated for adverse events.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Chemotherapy, Chemoradiotherapy, Surgery)
Number analyzed (Participants) | 81
percentage of participants | 72

ADVERSE EVENTS:
Arm/Group | Treatment (Chemotherapy, Chemoradiotherapy, Surgery)
Serious Adverse Events (participants affected / at risk) | 6/81
Other Adverse Events (participants affected / at risk) | 80/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Chemoradiotherapy, Surgery) (N=81)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (5)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 3 (4)
Disease progression (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (5)
Pain (General disorders) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 5 (5)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (4)
Platelet count decreased (Investigations) | 5 (6)
Weight loss (Investigations) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (2)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (4)
Dizziness (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Chemoradiotherapy, Surgery) (N=81)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 71 (190)
Hemolysis (Blood and lymphatic system disorders) | 2 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 2 (3)
Palpitations (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Ear disorder (Ear and labyrinth disorders) | 2 (5)
Hearing impaired (Ear and labyrinth disorders) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 9 (20)
Dry eye syndrome (Eye disorders) | 2 (2)
Eye disorder (Eye disorders) | 1 (1)
Flashing vision (Eye disorders) | 1 (2)
Vision blurred (Eye disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 14 (19)
Constipation (Gastrointestinal disorders) | 36 (65)
Diarrhea (Gastrointestinal disorders) | 38 (65)
Dyspepsia (Gastrointestinal disorders) | 7 (10)
Dysphagia (Gastrointestinal disorders) | 40 (87)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 6 (8)
Esophageal stenosis (Gastrointestinal disorders) | 2 (3)
Esophagitis (Gastrointestinal disorders) | 13 (15)
Flatulence (Gastrointestinal disorders) | 2 (5)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 18 (26)
Nausea (Gastrointestinal disorders) | 53 (106)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (3)
Salivary gland disorder (Gastrointestinal disorders) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (2)
Tooth development disorder (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 26 (38)
Chest pain (General disorders) | 5 (5)
Chills (General disorders) | 2 (3)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 60 (158)
Fever (General disorders) | 4 (4)
Hypothermia (General disorders) | 1 (1)
Pain (General disorders) | 7 (9)
Device related infection (Infections and infestations) | 1 (1)
Infective myositis (Infections and infestations) | 1 (1)
Paranasal sinus infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (3)
Upper respiratory infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (3)
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Injury, poisoning and procedural complications) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 5 (7)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 10 (16)
Alkaline phosphatase increased (Investigations) | 10 (16)
Aspartate aminotransferase increased (Investigations) | 6 (8)
Blood bilirubin increased (Investigations) | 3 (3)
Coagulopathy (Investigations) | 1 (1)
Creatinine increased (Investigations) | 5 (7)
INR increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (3)
Leukocyte count decreased (Investigations) | 70 (165)
Lymphocyte count decreased (Investigations) | 23 (44)
Neutrophil count decreased (Investigations) | 53 (112)
Platelet count decreased (Investigations) | 48 (88)
Weight gain (Investigations) | 2 (5)
Weight loss (Investigations) | 18 (27)
Anorexia (Metabolism and nutrition disorders) | 39 (67)
Blood glucose increased (Metabolism and nutrition disorders) | 37 (79)
Dehydration (Metabolism and nutrition disorders) | 27 (35)
Serum albumin decreased (Metabolism and nutrition disorders) | 18 (32)
Serum calcium decreased (Metabolism and nutrition disorders) | 15 (23)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 15 (24)
Serum magnesium increased (Metabolism and nutrition disorders) | 3 (4)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 10 (11)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (6)
Serum sodium decreased (Metabolism and nutrition disorders) | 28 (40)
Serum sodium increased (Metabolism and nutrition disorders) | 5 (7)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (10)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (6)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 10 (16)
Dysgeusia (Nervous system disorders) | 7 (13)
Headache (Nervous system disorders) | 10 (12)
Memory impairment (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 21 (48)
Syncope (Nervous system disorders) | 3 (6)
Tremor (Nervous system disorders) | 1 (3)
Anxiety (Psychiatric disorders) | 5 (8)
Confusion (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 10 (15)
Euphoria (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 19 (38)
Bladder pain (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (6)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (17)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 (22)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 30 (61)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (12)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 7 (9)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Hemorrhage (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (4)
Hypotension (Vascular disorders) | 6 (6)
Phlebitis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less